CLINICAL TRIAL: NCT00130156
Title: Effects of Combination Therapy With an α1-blocker (Sustained-release Preparation of Bunazosin or Doxazosin) in Inadequate Responders to an Angiotensin II Antagonist (Valsartan) in the Treatment of Patients With Mild to Moderate Essential Hypertension
Brief Title: Effects of Combination Therapy With Alpha-1 Blocker (Bunazosin or Doxazosin) in the Treatment of Patients With Mild to Moderate Essential Hypertension
Status: Completed | Phase: Phase 4 | Type: Interventional
Sponsor: Eisai Inc. (Industry)
Collaborators: Eisai Co., Ltd. (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: DTR-886-401
Record Dates: First submitted 2005-08-12; First posted 2005-08-15 (Estimated); Last update posted 2013-05-14 (Estimated); Status verified 2011-02

CONDITIONS: High Blood Pressure
Keywords: Blood pressure; SBP; DBP
MeSH Terms: conditions — Hypertension | interventions — bunazosin; Doxazosin; Valsartan

ARMS (2):
- 1 (Experimental)
  Interventions: Drug: Bunazosin; Drug: Valsartin
- 2 (Experimental)
  Interventions: Drug: Doxazosin; Drug: Valsartin

INTERVENTIONS:
Drug: Bunazosin — Patients will be randomized to the add-on treatment with Bunazosin (Detantol-R) 3 mg once-daily after breakfast for a total of eight weeks.
  Other Names: Detantol-R
  Arms: 1
Drug: Doxazosin — Patients will be randomized to the add-on treatment with Doxazosin (Doxaben XL) 4 mg once-daily after breakfast for a total of eight weeks.
  Other Names: Doxaben XL
  Arms: 2
Drug: Valsartin — After wash-out period, the eligible subjects will be treated with Valsartin (Diovan) 80 mg as the mono therapy for 5 weeks. If the blood pressures are inadequately responded, then the patients will be randomized to either Bunazosin (Detantol-R) or Doxazosin (Doxaben XL) along with Valsartin as the add-on treatment for 8 weeks.
  Other Names: Diovan

SUMMARY:
The purpose of this study is to investigate the efficacy and safety of Bunazosin with Valsartin compared to Doxazosin with Valsartin for patients with mild to moderate essential hypertension accompanied by metabolic syndrome.

DETAILED DESCRIPTION:
This clinical study will comprise a 1 to 2-week washout period, a 5-week mono therapy period with AngiotensinⅡantagonist, and an 8-week alpha blocker add-on treatment period. Total study period will be 15 weeks.

ELIGIBILITY:
Inclusion Criteria:

Subjects with mild to moderate essential hypertension, with the following criteria:

1. Washout period (Week -2)

   * Male or female subjects aged 20 to 80 years
   * Systolic blood pressure (SBP):140 mm Hg but <180 mm Hg and/or diastolic blood pressure (DBP):90 mm Hg but <110 mm Hg
   * Subjects who have given written informed consent prior to participation in the trial and who undertake to comply with the protocol
2. Angiotensin II antagonist mono-therapy period (week 0)

   * Subjects with systolic blood pressure >= 140 mm Hg but <180 mm Hg and/or diastolic blood pressure >= 90 mm Hg but <110 mm Hg
   * Presence of any 2 of the following 4 risk factors
   * Waist circumference: male > 90 cm, female > 80 cm
   * Triglycerides >= 150 mg/dl
   * HDL cholesterol: male < 40 mg/dl, female < 50 mg/dl
   * Fasting glucose >= 110 mg/dl
3. Angiotensin II antagonist with add-on Bunazosin or Doxazosin treatment period (Week 5)

   * SBP >=140 mm Hg or decrease < 10 % OR
   * DBP >=90 mm Hg or decrease < 10 % comparing the blood pressure at the entry of the Angiotensin II antagonist mono-therapy period.

Exclusion Criteria:

Subjects with the following conditions are not eligible for participation：

a) Washout period (Week -1 or -2)

* Subjects with severe hypertension (SBP>=180 mm Hg or DBP>=110 mm Hg).
* Subjects who have proven or suspected hypersensitivity to quinazoline derivatives
* Subjects who have a history of alcohol or drug abuse.
* Subjects with past or present evidence of cancer
* Subjects who have a past history of arterial fibrillation, heart failure (LVEF<40%), acute coronary syndrome, myocardial infarction, stroke or severe arrhythmia.
* Subjects who are severely obese (BMI>30 kg/m2)
* Women who are pregnant or lactating or suspected of being pregnant.
* Subjects who have previously participated in any clinical trial of new or unapproved substances within the 12 weeks before starting of washout period
* Subjects on other anti-hypertensive or lipid-lowering medication
* Inability to return for scheduled visits or comply with any other aspect of the Protocol
* Subjects with poorly controlled diabetes mellitus (HbA1c > 10%)
* Subjects with concurrent serious hepatic or renal disorders (defined as AST and/or ALT > 3 times upper normal limit or Cr > 2mg/dl).
* Subjects who, in the opinion of the investigators, are poor medical candidates or pose any other risk for therapy with an investigational drug.

Ages: 20 Years to 80 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 93 (Actual)
Dates: Start 2005-10; Primary Completion 2008-09 (Actual); Study Completion 2009-03 (Actual)

PRIMARY OUTCOMES:
Blood Pressure | Week 0, Week 4, Week 9, Week 13.

SECONDARY OUTCOMES:
Safety and tolerability. | Week 4, Week 9, Week 13.

CONTACTS AND LOCATIONS:
Overall Officials: Ya-hui Cheng, Study Director — Medical Affairs Department , Eisai Taiwan Inc.
Locations (1):
- National Taiwan University Hospital., Taipei, Taiwan